CLINICAL TRIAL: NCT06965322
Title: Prospective Observational Study on the Detection of Pleuropulmonary Manifestations in Rheumatoid Arthritis
Brief Title: Study on the Detection of Pleuropulmonary Manifestations in Rheumatoid Arthritis
Acronym: REASSESS
Status: Recruiting | Type: Observational
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Other Study IDs: EK Nr: 1086/2024
Record Dates: First submitted 2024-11-11; First posted 2025-05-11 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Rheumatic Arthritis; Interstitial Lung Disease in Patients With Rheumatoid Arthritis
Keywords: rheumatoid arthritis; interstitial lung disease; risk prediction; RA-ILD
MeSH Terms: conditions — Rheumatic Fever; Arthritis, Rheumatoid; Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood sample collection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to develop a standardized, risk-adapted screening protocol for detecting pleuropulmonary manifestations in patients with rheumatoid arthritis. To assess the risk of these manifestations, a comprehensive range of functional and clinical evaluations will be performed and correlated with structural lung assessments using computed tomography (CT).

DETAILED DESCRIPTION:
The objective of the study is the establishment of a standardized risk-adapted screening protocol for detecting pleuropulmonary manifestations in patients with rheumatoid arthritis. To determine the risk of pleuropulmonary manifestation in RA, clinical (pulmonological and rheumatological specialist examination including standardized disease activity and symptom scores), laboratory (e.g. RF, ACPA, CRP, CEA), lung function (incl. body plethysmography, TLCO, FeNO, SMWT), sonographic (thoracic ultrasound, joint ultrasound), and demographic (e.g., age, gender) factors will be considered. A machine learning (ML) based risk-modeling approach will be utilized to create the screening tool. For further external validation and clinical application, a freely accessible online tool and a mobile app will be developed based on the existing model.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years diagnosed with rheumatoid arthritis according to current ACR/EULAR criteria
* Residence in Austria
* Signed and dated consent of the patient in accordance with ICH-GCP guidelines

Exclusion Criteria:

* pregnancy
* age below 18 years
* Contraindications to study-related routine examinations (e.g., inability to draw blood due to needle phobia, no CT scan possible due to claustrophobia, pregnancy, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years or older, currently residing in Austria, diagnosed with rheumatoid arthritis according to the current ACR/EULAR criteria, will be eligible for study entry.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2028-05-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of RA patients with pleuropulmonary involvement according to an AI-supported multiparametric risk profile analysis | single point (baseline)
  AI-supported risk factor-based analysis of pleuropulmonary involvement in RA patients assessed at a single time-point (baseline assessment). A multiparametric AI-supported evaluation based on clinical, sonographic, pulmonary function, laboratory, and exercise performance tests defines an RA population at high risk for the presence of pleuropulmonary involvement.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Innsbruck, Innsbruck, Austria, Austria

IPD SHARING:
Plan to Share IPD: Undecided